CLINICAL TRIAL: NCT03275272
Title: Effect of maternalBMI and Type of Infants Feeding on IGF-1in Infants as Early Marker of Childand Adult Hood Obesity
Brief Title: Effect of Maternal BMI and Type of Infants Feeding on IGF-1 in Infant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, N M Shahata, Nesma Mohamed Ezz ElDien Shahata, Assiut University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IGF-1level in infants
Record Dates: First submitted 2017-09-06; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: IGF1 Deficiency
MeSH Terms: conditions — Insulin-Like Growth Factor I Deficiency

STUDY DESIGN:
Intervention Model Description: Measurment of maternal BMI and serum level if IGF-1 in infant
Masking Description: Measurment of blood level of IGF-1 and Maternal BMI
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- level of IGF-1 in infant (Other): Measurment of blood level of IGF-1 In infants
  Interventions: Diagnostic Test: level of IGF-1 in infants

INTERVENTIONS:
Diagnostic Test: level of IGF-1 in infants — Measurment of blood level of IGF-1 in infants

SUMMARY:
IGF-I is a mitogenic and antiapoptotic. paracrine growth factor expressed in all fetal organ. and is essential in fetal and neonatal growth, differentiation and development Several lines of evidence suggest that IGF-I levels are associated with birth weight -furthermore higher IGF-I levels are associated with higher BW, but not with lower birth weight]. In adulthood, elevated concentrations of IGF-I are associated with an increased risk of obesity and many cancers, including breast, lung, head and neck, colorectal, pancreas, synovial sarcoma, and prostate canc. Although concentrations of circulating IGF-I levels vary considerably by race/ethnicity and maternal pre-pregnancy obesity, few studies included African American women an ethnic group that has an almost 9% higher BMI than European-American women

DETAILED DESCRIPTION:
For healthy mother ,breastfeeding represent the gold standard for infant health, and infant formula development aims at mimicking the physiological response to human milk intake. while protein content is essential to promote growth and brain development, protein intakes in late infancy have been found to be quite high and to exceed required intakes by large margins )Ohlund and ,Hernell , 2010)

More over ,high protein intake was associated with increased weight gain and higher adiposity in infancy and child hood )Singhal and kennedy , 2010 ) further more, protein intake of breast-fed infant is generally lowerand may relate to lower risk of obesity later in life)Harder and Betgmann , 2005 )

one potential mechanism involves an enhanced stimulation of the secretion of Insulin growth factor(IGF-1)strophic hormone involved in longitudinal growth as well as muscle and fat mass development (Rolland et el,1995 )

• General research statement and Justification of the research

A-Maternal BMI and IGF-1 level in infants There's a positive association among term infant with elevated IGF-1 level and increased risk with higher birthweight. This positive association most apparent in infant born to obese women PubMed).

Maternal obesity is rising with subsequent increase risk of childhood obesity offspring of overweight and obese women (whit Take ,2004 )

Obese women have difficulties in initiating and maintaining breastfeeding because of defects in their hormonal response to suckling. (Rasmussen and kjolhede , 2004 )

B-Type of Feeding And IGF-1 level in infant Breastfed infant tend to be smaller and have lower endogenous production of IGF-1 than formula fed infant this attributed to their higher protein content of formula(SOCHA ET Al2011) how ever this relation reverse as childhood progress at age 17 young adult hood who has breastfed had higher IGF-1) than the formula fed (LANKAERET Al 2009) Large Danish birth cohort reported that IGF-1 concentration at age 3month were higher in formula feeding infants than in breastfeeding infants (CHellakooty et al., 2006 ).

Nutritional view on breast feeding Posted on July 14, 2013 by Thomas Sherman

C-Relationship between IGF-1 and Childhood obesity and adulthood obesity. Rapid growth in infancy is associated with later over weight and obesity Faster weight gain during infancy is associated with increased risk of subsequent obesity and related metabolic traits (Longitudinal birth cohort study and analysis pediatr Res 2002;52:863-7)

ELIGIBILITY:
Inclusion Criteria:

* infants from two to three month and thier mother

Exclusion Criteria:

* 1 -VLBW. 2-preterm infants. 3-IUGR 4-mother with hormonal disturbance

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
IGF-1 level in infants | One year
  Effect of maternal BMI and type of feeding of infants on IGF-1on infants

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hansen-Pupp I, Lofqvist C, Polberger S, Niklasson A, Fellman V, Hellstrom A, Ley D. Influence of insulin-like growth factor I and nutrition during phases of postnatal growth in very preterm infants. Pediatr Res. 2011 May;69(5 Pt 1):448-53. doi: 10.1203/PDR.0b013e3182115000. PMID 21263374
- [Result] Lineham JD, Smith RM, Dahlenburg GW, King RA, Haslam RR, Stuart MC, Faull L. Circulating insulin-like growth factor I levels in newborn premature and full-term infants followed longitudinally. Early Hum Dev. 1986 Feb;13(1):37-46. doi: 10.1016/0378-3782(86)90096-4. PMID 3956421
- [Result] Hikino S, Ihara K, Yamamoto J, Takahata Y, Nakayama H, Kinukawa N, Narazaki Y, Hara T. Physical growth and retinopathy in preterm infants: involvement of IGF-I and GH. Pediatr Res. 2001 Dec;50(6):732-6. doi: 10.1203/00006450-200112000-00017. PMID 11726732